CLINICAL TRIAL: NCT05807984
Title: A Prospective Phase II Clinical Study of Carbon Ion Re-irradiation in Unresectable Locally Recurrent Rectal Cancer
Brief Title: Re-irradiation Therapy of Locally Recurrent Rectal Cancer With Carbon Ion
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xin Cai (Other)
Responsible Party: Sponsor-Investigator, Xin Cai, Deputy chief physician, Shanghai Proton and Heavy Ion Center
Organization: Shanghai Proton and Heavy Ion Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-CRC2021-01
Record Dates: First submitted 2023-02-16; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Rectal Cancer; Recurrent
MeSH Terms: conditions — Rectal Neoplasms; Recurrence

STUDY DESIGN:
Intervention Model Description: carbon ion therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- carbon ion therapy for unresectable local recurrent rectal cancer (Experimental)
  Interventions: Radiation: Carbon ion radiation therapy DT: 74Gy/20 fractions

INTERVENTIONS:
Radiation: Carbon ion radiation therapy DT: 74Gy/20 fractions — patients with unresectable local recurrent rectal cancer will be treated with carbon ion radiation therapy as re-irradiation

SUMMARY:
Prospective phase II clinical study aim to explore the clinical outcome of patients with unresectable locally recurrent rectal cancer (LRRC) treated with re-irradiation by carbon ion radiotherapy (CIRT)

ELIGIBILITY:
Inclusion Criteria:

* 1) pathologically confirmed rectal adenocarcinoma (including mucinous adenocarcinoma and signet-ring cell carcinoma) and LRRC confirmed by biopsy or clinical diagnosis,
* 2) received a radical operation for their primary tumor and regional lymph nodes,
* 3) received chemo-radiation or radiation in pelvic before CIRT,
* 4) received re-irradiation by CIRT after their pelvic radiotherapy.

Exclusion Criteria:

* 1) received more than once prior radiotherapy in the same treatment field,
* 2) time to the last radiotherapy was <1 year,
* 3) space between the lesion to organ at risk (OARs) (bladder or digestive tract) was too close (<5 mm).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
local control | Local control at 3 years after CIRT
  local control rate of the lesion treated by CIRT

SECONDARY OUTCOMES:
overall survival | 3 years after CIRT or patient died, measured erery 3 months after CIRT
  survival rate after CIRT
progression free survival | 3 years after CIRT or patient died, measured erery 3 months after CIRT
  progression free survival rate after CIRT

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy ion center, Shanghai, Pudong, China

IPD SHARING:
Plan to Share IPD: No